CLINICAL TRIAL: NCT05955040
Title: Treatment of Elevated Blood Pressures in Early Pregnancy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study has closed due to difficulty in enrollment.
Sponsor: Marshall University (Other)
Responsible Party: Principal Investigator, Jesse Cottrell, Assistant Professor of Maternal Fetal Medicine, Marshall University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1889318
Record Dates: First submitted 2023-06-01; First posted 2023-07-20 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Elevated Blood Pressure; Pregnancy Induced Hypertension
MeSH Terms: conditions — Hypertension; Hypertension, Pregnancy-Induced | interventions — Nifedipine; Labetalol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): Treatment of elevated blood pressures (120 or greater systolic OR 80 or greater diastolic)
  Interventions: Drug: Nifedipine; Drug: Labetalol
- Non-treatment Group (No Intervention): Non-treatment of blood pressures between 120-139 systolic and 80-89 diastolic

INTERVENTIONS:
Drug: Nifedipine — Standard of care for treatment of elevated blood pressure during pregnancy
  Arms: Treatment Group
Drug: Labetalol — Standard of care for treatment of elevated blood pressure during pregnancy
  Arms: Treatment Group

SUMMARY:
This is a randomized controlled trial comparing the outcomes of treatment and non-treatment of elevated blood pressures in early pregnancy.

DETAILED DESCRIPTION:
Patients will be randomized to treatment of elevated blood pressures (120 or greater systolic OR 80 or greater diastolic) versus non-treatment. After randomization to treatment, patient's will be treated with either nifedipine or labetalol (both medications that are standard of care for treatment of elevated blood pressure during pregnancy).

The purpose of this study is two-fold: 1) Determine if treatment of elevated blood pressures (120 or greater systolic OR 80 or greater diastolic) versus non-treatment improves maternal and fetal outcomes and 2) determine if ICG directed treatment is optimal as ICG will not be used to determine treatment medication (this will be done by secondary analysis after conclusion of the study).

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for obstetric care at Marshall University (Huntington office and Teays Valley office) between 12 and 16 weeks gestation with a systolic blood pressure of 120 or greater OR a diastolic blood pressure of 80 or greater. Eligibility for this study will be have blood pressures between 120-139 systolic and 80-89 diastolic. Randomization to control, labetalol, or nifedipine will be performed after patient consent.

Exclusion Criteria:

* Patients already be on medication for hypertension.
* Patients with the diagnosis of chronic hypertension
* Patients with a BP of 140 or greater systolic OR 90 or greater diastolic (this meets criteria for chronic hypertension in pregnancy).
* Patients actively using any illicit substance or have history of substance use disorder.
* Patients who are actively consuming alcohol during pregnancy.
* Patients with Type I or Type II Diabetes Mellitus.
* Patients with end stage renal disease.
* Patients less then 12 weeks gestation or greater than 16 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 2 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Treatment of elevated blood pressures | through study completion, an average of 1 year
  Patient age
Treatment of elevated blood pressures | through study completion, an average of 1 year
  BMI
Treatment of elevated blood pressures | through study completion, an average of 1 year
  delivery weeks
Treatment of elevated blood pressures | through study completion, an average of 1 year
  systemic vascular resistance
Treatment of elevated blood pressures | through study completion, an average of 1 year
  heart rate
Treatment of elevated blood pressures | through study completion, an average of 1 year
  blood pressure
Treatment of elevated blood pressures | through study completion, an average of 1 year
  gravidity
Treatment of elevated blood pressures | through study completion, an average of 1 year
  parity
Treatment of elevated blood pressures | through study completion, an average of 1 year
  abortions
Treatment of elevated blood pressures | through study completion, an average of 1 year
  gestational hypertension
Treatment of elevated blood pressures | through study completion, an average of 1 year
  inhouse days
Treatment of elevated blood pressures | through study completion, an average of 1 year
  preeclampsia
Treatment of elevated blood pressures | through study completion, an average of 1 year
  birth weight percentile
Treatment of elevated blood pressures | through study completion, an average of 1 year
  Apgar 1 min
Treatment of elevated blood pressures | through study completion, an average of 1 year
  Apgar 5 min
Treatment of elevated blood pressures | through study completion, an average of 1 year
  NICU days

SECONDARY OUTCOMES:
ICG directed treatment | through study completion, an average of 1 year
  Compare cardiac output
ICG directed treatment | through study completion, an average of 1 year
  mean arterial pressure
ICG directed treatment | through study completion, an average of 1 year
  systemic vascular resistance among groups treated with nifedipine, labetalol, and the control group

CONTACTS AND LOCATIONS:
Locations (1):
- Marshall Obstetrics and Gynecology, Huntington, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided